CLINICAL TRIAL: NCT06098521
Title: Project CONSENT: a Randomized Controlled Trial to Evaluate Cognitive Behavioral Therapy for the Prevention of Sexual Recidivism
Brief Title: Project CONSENT: Cognitive Behavioral Therapy to Prevent Sexual Recidivism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Prison and Probation Services (Unknown)
Responsible Party: Principal Investigator, Christoffer Rahm, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-04498-01
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Sexual Offending Behavior
Keywords: Sexual Offending; Recidivism; Cognitive behavioral therapy; Randomized controlled trial
MeSH Terms: conditions — Recidivism | interventions — Consent Forms

STUDY DESIGN:
Intervention Model Description: A randomized waiting list controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONSENT and Follow-up (Experimental): The therapy in the CONSENT program will be delivered twice a week (total time 12 ± 2 weeks), with measurement after 16±2 weeks. Participants in this arm will have a follow-up period of 16±2 weeks.
  Interventions: Behavioral: CONSENT
- Waiting list and CONSENT (Experimental): Participants will be on waiting list for 16±2 weeks. After waiting list participants are offered the CONSENT program including therapy delivered twice a week (total time 12 ± 2 weeks), with measurement after for 16±2 weeks.
  Interventions: Behavioral: CONSENT

INTERVENTIONS:
Behavioral: CONSENT — The CONSENT program is a risk-, need- and responsivity (RNR) based CBT program primarily focused on reducing risk of sexual reoffending, that consists of 18-26 one-to-one sessions in correctional settings.

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of cognitive behavioral therapy (CBT) on sexual recidivism risk in a Swedish sample of incarcerated men convicted of sexual offenses. The main question it aims to answer is: Does the CBT program CONSENT reduce the risk of recidivism in sexual offenses among males convicted of sexual offending? The CONSENT program, specifically targeting risk factors for sexual recidivism, will be compared with a waiting list. The evaluation will focus on potential change in dynamic risk factors for sexual recidivism. The study is part of the project Preventing Sexual Abuse: CBT Programs for Convicted Men and Women in a Correctional Setting.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the short-term effects of the CONSENT program. To improve participation and responsivity and minimize any unintentional side effects, men's experiences of CONSENT are also sought.

Firstly, clients' changes will be examined in two complementary ways: through professionals' assessments and through clients' assessments using questionnaires. Secondly, changes in risk will be examined at two time points (after the program and at the 4-month follow-up), and the willingness to change in order to obtain additional complementary measures of the intended change process.

The primary research question and hypothesis, based on professionals' assessment (assessment not made by the same person conducting the program), is as follows:

1. Does the CONSENT program reduce the risk of recidivism in sexual offenses, as assessed by professionals, among males convicted of sexual offending (initially assessed as having a moderate risk of sexual offense recidivism)? The main hypothesis is that the estimated risk of recidivism in sexual offenses will be reduced more among men participating in CONSENT than among men on the waiting list, based on professionals' assessments.

   The following secondary research questions complement the primary question:
2. Does social problem-solving change during participation in CONSENT?
3. Does emotional self-regulation change during participation in CONSENT?
4. Does the willingness to change among participants in CONSENT change?
5. What changes are sustained at the four-month follow-up assessment?
6. Does self-reported risk of committing sexual offenses against children change during participation in CONSENT?
7. Do sexual urges involving children change during participation in CONSENT?

Participants will also report any negative side effects and serious adverse events resulting from participating in CONSENT, as well as describe positive and negative experiences related to their participation. Please note that research questions 5 and 6 apply only to individuals convicted of sexual offenses against children and/or who indicate a sexual interest in children in the LASSIE instrument measuring paraphilic interests.

The trial will be conducted within the Swedish Prison and Probation Service at prisons specialized in individuals convicted of sexual offending.

ELIGIBILITY:
The study population is a subgroup of the study population in another study within the same project. Eligibility criteria for that study:

Inclusion Criteria:

* Men aged 18 and above sentenced to imprisonment within the Swedish Prison and Probation Service.
* and offense falls under Chapter 6 of the Swedish Penal Code concerning sexual offenses or relates to child pornography offenses.
* and risk of recidivism for sexual offenses is assessed as "average" or higher according to the Risk Matrix 2000.
* and provided signed informed consent.

Exclusion Criteria:

* Individuals with apparent influence at the time of assessment due to severe psychiatric conditions such as pronounced psychotic symptoms or dementia.
* or difficulties conducting interviews and self-assessments/surveys due to language barriers in understanding the Swedish language.
* or difficulties in fully understanding the conditions for consenting to participate.

Additional eligibility criteria for the current trial:

Inclusion Criteria

* Inclusion criteria for Consent are met:
* and the risk of relapse in sexual offenses is assessed as average risk of relapse in sexual offenses with Risk Matrix 2000
* and the participant does not meet the inclusion criteria for SEIF (medium to high risk of relapse in sexual offenses and concurrent paraphilia and/or sexual preoccupation and/or emotional identification with children and/or extensive responsivity issues).
* and a total score (all items included) on The Sex Offender Treatment Intervention and Progress Scale (SOTIPS) of ≤20
* and ≥9 months to halftime of sentence, when it becomes possible to apply for reintegration measures (including 12±2 weeks in the program and 4 weeks without the program, 16±2 weeks on the waitlist/follow-up, and time for assessment and inclusion) or ≥9 months left until conditional release and special conditions that state that reintegration measures are not allowed.
* and written informed consent.

Exclusion Criteria

- Any exclusion criteria for Consent are met: difficulties in understanding the program's content and carrying it out due to difficulties in understanding the Swedish language

* or severe or ongoing unstable psychiatric conditions or other conditions that hinder participation (high suicide risk, significant psychotic symptoms, diagnosed intellectual disability, or other serious cognitive illness such as dementia)
* or ongoing participation in another psychological program. If potential research subjects have other programs in their sentence plan, participation in the study will be prioritized if it is deemed appropriate in individual cases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in The Sex Offender Treatment Intervention and Progress Scale (SOTIPS) score, a sum score based on a 11 selected items. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  A risk/need measurement based on the SOTIPS assessment, limited to a summation measure (0-33 points; higher scores indicate higher risk) based on the following items: Sexual Offense Responsibility, Sexual Attitudes, Sexual Risk Management, Criminal Rule-Breaking Behavior, Criminal Rule-Breaking Attitudes, Stage of Change, Cooperation with Treatment, Emotional Management, Problem Solving, Impulsivity, and Social Influence.

SECONDARY OUTCOMES:
Change in central criminogenic needs, i.e., social problem-solving ability and emotion regulation skills. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  Measured with the Social Problem Solving Inventory-Revised (SPSI-R) (25-125 points, higher scores indicate more difficulties).
Change in central criminogenic needs, i.e., social problem-solving ability and emotion regulation skills. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  Measured with the Emotion Regulation Scale-Brief version (DERS-16)(16-80 points; higher scores indicate more difficulties).
Motivation for change. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  Measured with The Change Questionnaire (TCQ)(0-30 points, higher scores indicate more motivation).
Change in sexual urges involving children. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  Measured by Sexual Symptom Assessment Scale (SASS)(0-48 points; higher scores indicate more urges). This outcome is only for the subgroup that is convicted of a child sexual offence or self-report a sexual interest in children.
Change in self-reported risk. | 1) Pre-measurement at baseline. 2) Post-measurement after waiting list / CONSENT (16±2 weeks). 3) Post-measurement after CONSENT/Follow-up (16±2 weeks).
  Measured with a version of the Sexual Child Molestation Risk Assessment (SChiMRA) (visual analogue scale 0-10, higher points indicate higher risk). Each of the three items are reported separately. This outcome is only for the subgroup that is convicted of a child sexual offence or self-report a sexual interest in children.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Rahm, M.D., Ph.D., Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm, Stockholm County
  - Swedish Prison and Probation Service, Norrköping

IPD SHARING:
Plan to Share IPD: No